CLINICAL TRIAL: NCT05459506
Title: Investigating the Relationship Between Development of Autoimmunity Due to Severe Acute Respiratory Syndrome (SARS)-Corona Virus-2 (CoV2) Infection and Long-term Health Post Recovery
Brief Title: Investigating Development of Autoimmunity in Post-Acute COVID-19 Syndrome (PACS)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Other Study IDs: COV-IMM001
Record Dates: First submitted 2022-07-13; First posted 2022-07-15 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: COVID-19 Pandemic
Keywords: Post Acute Sequelae; Long Covid; Rheumatology; Auto Immune
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and sputum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects with Post Acute Sequale SARS-CoV-2 (PSAC): Participants with PASC
- Subjects with COVID but not PASC: Subjects confirmed COVID-19 positive without Post Acute Sequale SARS-CoV-2 (PASC)

SUMMARY:
The coronavirus pandemic has severely affected healthcare systems and changed life as everyone know it, globally. Apart from the acute phase disease complications, it is now apparent that a significant proportion (15%) of patients who recover continue experiencing symptoms such as chronic fatigue, shortness of breath, joint pains, cognitive impairment ("brain fog"), etc. for several months, if not for life. This syndrome has been labeled as "long-COVID" or Post-Acute COVID-19 Syndrome (PACS) and can happen to anyone whether you're young, old, healthy, or have a chronic illness. One can get it even if the COVID-19 symptoms were mild. There is no confirmed cause as to why this happens. However, there is data to support that inappropriate activation of the immune system by the virus may play a role. While our immune system is programmed to protect us against foreign invaders (such as viruses), in this case, it is directed against elements of our own. The net result is autoimmunity, where the immune system produces autoantibodies that cause damage to the body. This may lead to the development of chronic and serious diseases like lupus, rheumatoid arthritis, vasculitis, scleroderma, and others.The aim of our study is to understand the exact impairment of the immune system, why these patients develop autoantibodies, characterize their impact on the clinical symptoms of PACS, and, potentially, identify ways to modify this. The study's impact is significant since it is projected that 150000 Canadians will experience (or are already experiencing) this syndrome.

DETAILED DESCRIPTION:
Background: As of April 10th, 2021, >1 million Canadians have contracted Coronavirus-2019-disease (COVID-19), with 398,835 infected in Ontario of whom 92% are deemed "recovered" by public health. Despite the recovery, a considerable section (10-15%) of COVID-19 survivors, irrespective of their severity (hospitalized or mild), continue to have symptoms or develop new ones. These vary in type and severity between individuals, ranging chronic fatigue, anosmia, dyspnea, diffuse pain, anxiety, cognitive impairment that is not attributed to any clinical diagnosis. This is now termed the Post-Acute COVID-19 Syndrome (PACS) or long-COVID. Much remains unknown as to what underlies this constellation of symptoms and what more severe pathologies it can lead to.

Rationale to study autoimmunity in PACS: First, diverse circulating auto antibodies and lymphopenia are associated with COVID-19 severity. Second, though the male: female sex ratio for contracting the infection and recovery rate is comparable, recent studies indicate PACS to be more prevalent in females, with increasing age and BMI. Taken together these are hallmark etiological factors and demographics underlying diverse autoimmune pathologies. Third, the lung being the primary affected organ may be the site of chronic auto inflammation itself. There is evidence of auto reactivity and detectable autoantibodies in sputa associated with autoimmune diseases with pulmonary complications (such as rheumatoid arthritis, vasculitis). Finally, there is a growing body of anecdotal evidence highlighting autoimmune diagnoses post-COVID, ranging from Guillain Barre to vasculitis to lupus, in otherwise previously healthy individuals. Our preliminary data suggests 35% of individuals post-COVID have >2 circulating autoantibodies at a high disease-modifying titre, significantly associated with health outcomes. While viruses, in general, have the innate capacity to induce autoimmunity (may not be specific to SARS-CoV2), the magnitude of PACS individuals affected warrants further investigation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years up
* Positive PCR or antibody test
* 12 weeks post acute Covid infection with PASC

Exclusion Criteria:

* Pre-existing Auto- immune disease
* Chronic/ secondary infections
* Active Neoplasm
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Confirmed COVID diagnosis by PCR/sero-positive based and deemed recovered by public health.
  A control age-sex matched population who had symptoms (infection) and tested negative for SARS-CoV2 with a PCR test, will be recruited.
  A control age-sex matched population (n=20) with no infection within 4 weeks of recruitment or ever tested positive for COVID and with no known medical conditions and a non-significant smoking history (less than ten years of smoking history).
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-06-25 (Actual); Primary Completion 2024-03-25 (Estimated); Study Completion 2024-03-25 (Estimated)

PRIMARY OUTCOMES:
Development of auto antibodies (in blood and/or sputum) in PACS and a clinical diagnosis of an autoimmune condition over time . | Baseline to 18 months
  Detection of autoantibodies in PASC and a clinical diagnosis of an autoimmune condition over time .

CONTACTS AND LOCATIONS:
Overall Officials: Manali Mukherjee, PhD, Principal Investigator — McMaster University
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No